CLINICAL TRIAL: NCT02088983
Title: Effects of CDP-Choline on Gating and Cognitive Deficits in First Episode Schizophrenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Dr. Verner Knott, Director, Clinical Neuroelectrophysiology and Cognitive Research Laboratory, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2013031
Record Dates: First submitted 2014-03-12; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: First Episode Schizophrenia
MeSH Terms: interventions — Cytidine Diphosphate Choline; Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- CDP-Choline (Experimental): Single dose of 500 mg, 1000 mg, or 2000 mg given in one of 4 test sessions
  Interventions: Dietary Supplement: CDP-Choline
- Placebo (cellulose) (Placebo Comparator): Given randomly in one of the 4 testing sessions as a comparison
  Interventions: Dietary Supplement: Cellulose

INTERVENTIONS:
Dietary Supplement: CDP-Choline — Capsule
  Other Names: citicoline
  Arms: CDP-Choline
Dietary Supplement: Cellulose — Capsule
  Arms: Placebo (cellulose)

SUMMARY:
People with schizophrenia tend to have problems with attention and concentration. Studies found that these patients are unable to block or gate out non-relevant and distracting information (e.g., noises). This may lead to brain overload. Cognitive abilities like concentration, memory, and learning may worsen. This ability to filter sensory information has been linked to a gene that affects the way nicotine acts in the brain. Patients with schizophrenia have a high rate of cigarette smoking. 60% to 90% smoke compared with 25% of the general population. It has been suggested that these patients may use nicotine to improve their ability to block out distracting information. Brain wave activity (EEG) in response to sounds has been proved useful in understanding this gating problem. The present study uses EEG measures and performance tasks to find out what a new nicotine-like treatment, which will be added to ongoing treatment medications, does to gating and cognition. It is hoped that this new treatment will improve the way in which patients process information, as this may help them in day-to-day activities.

DETAILED DESCRIPTION:
* A sample of 40 patients will be recruited from the Champlain First Episode Psychosis Program, a service of The Ottawa Hospital, which is run in conjunction with the Schizophrenia Program of the Royal Ottawa Mental Health Center.
* In this randomized, double-blind, placebo-controlled, cross-over design study, participants will attend the laboratory for four test sessions and will receive either a single dose of CDP-choline (500 mg, 1000 mg or 2000 mg) or placebo at each test session
* EEG recordings (with a focus on the P50 ERP) and cognitive testing measures will be collected in each test session to determine any possible gating or cognitive effects of CDP-choline. A saliva sample will also be collected to determine any genetic differences in the effects of CDP-choline
* The investigators carefully engineered study aims to assess the optimal dosing of a nicotinic cholinergic agonist, CDP-choline to increase P50 suppression and cognitive efficacy in an early schizophrenia population with abnormal P50 suppression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 - 60 years old
* Meet DSM-IV/DSM-IV-TR criteria for First Episode Schizophrenia
* Clinical stability of the past 2 months [assessed with the PANSS]
* Treatment with a single antipsychotic medication (concomitant psychiatric medications allowing on an "if needed basis".
* Smoker or non-smoker

Exclusion Criteria:

* Any comorbid Axis I disorder including a current or recent history of alcohol/substance abuse
* A clinically significant medical illness or organic brain disorder known to cause psychosis or cognitive impairment
* Recent head trauma (<6mos)
* Major learning disability
* Body mass index >38kg/m¬2
* Use of illicit drugs
* Abnormal hearing

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Acute Effects of CDP-Choline | 1 year
  To examine the acute effects of CDP-choline on P50 auditory gating deficits in FES. Complementing this, we will measure CDP-choline response as a function of dose, administering doses at 3 clinically recommended levels (500 mg, 1000 mg, 2000 mg).

SECONDARY OUTCOMES:
Acute Effects of CDP-Choline on Cognition | 1 year
  Although sensory processing and neurocognitive processing show poor interrelatedness in SZ (vs. healthy controls) and evidence supporting a relationship between sensory gating and specific cognitive domains is mixed, auditory gating consistently predicts variance in tasks of attention, working memory and less so in executive functioning. Its nicotinic improvements in relatively low-level sensory processes might also be expected to translate into benefits for more complex cognitive processes that are required for functional daily living. A secondary objective of this research will assess the acute effects of CDP-choline on cognitive operations. This will be conducted using a test battery assessing seven orthogonal domains of cognition designated by MATRICS as targets for clinical assessment of potential cognitive enhancers for SZ.

OTHER OUTCOMES:
Exploratory Objective: Genetic Differences | 1 year
  Although the sample size is relatively small, this study will begin to explore differences in CDP-choline response by classifying patients by CHRNA7 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Verner Knott, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa Institute of Mental Health Research, Ottawa, Ontario, Canada